CLINICAL TRIAL: NCT03650608
Title: A Dose Block-randomized, Double-blind, Placebo Controlled, Dose-escalation Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics After Single Dosing of HL217 Eye Drop in Healthy Male Subjects
Brief Title: A Clinical Trial to Evaluate Tolerability and Pharmacokinetics of HL217 Eye Drop in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: HL217-101
Record Dates: First submitted 2018-06-19; First posted 2018-08-29 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2018-08

CONDITIONS: Healthy Subject

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Cohort 1: HL217 Ophathalmic Solution QD (Experimental): HL217 3mg/mL, Ophthalmic solution, two drop once a day
  Interventions: Drug: Cohort 1: HL217 Ophathalmic Solution QD
- Cohort 2: HL217 Ophathalmic Solution BID (Experimental): HL217 3mg/mL, Ophthalmic solution, two drop twice a day
  Interventions: Drug: Cohort 2: HL217 Ophathalmic Solution BID
- Cohort 3: HL217 Ophthalmic Solution QID (Experimental): HL217 3mg/mL, Ophthalmic solution, two drop four times a day
  Interventions: Drug: Cohort 3: HL217 Ophthalmic Solution QID
- Placebo Ophthalmic solution (Placebo Comparator): Placebo Ophthalmic solution, two drop once or twice or four times a day
  Interventions: Drug: Placebo Ophthalmic solution

INTERVENTIONS:
Drug: Cohort 1: HL217 Ophathalmic Solution QD — Cohort 1 (Once a day)
  Other Names: 3mg/mL
  Arms: Cohort 1: HL217 Ophathalmic Solution QD
Drug: Cohort 2: HL217 Ophathalmic Solution BID — Cohort 2 (Twice a day)
  Other Names: 3mg/mL
  Arms: Cohort 2: HL217 Ophathalmic Solution BID
Drug: Cohort 3: HL217 Ophthalmic Solution QID — Cohort 3 (Four times a day)
  Other Names: 3mg/mL
  Arms: Cohort 3: HL217 Ophthalmic Solution QID
Drug: Placebo Ophthalmic solution — Placebo
  Other Names: Placebo
  Arms: Placebo Ophthalmic solution

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and PK parameters in healthy subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability and PK parameters of HL217 after single eye drop administration at different doses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject, aged between 18 and 50 years inclusive
2. Non-smoker subject or smoker of not more than 10 cigarettes a day and able to stop smoking 24 hour prior to admission until discharge
3. Body weight ≥ 50 kg and BMI between 18 and 30 kg/m²
4. Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination) including complete ocular examination
5. Normal Blood Pressure (BP) and Heart Rate (HR) after 10 minutes in supine position:

   * 90 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 140 mmHg
   * 45 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 90 mmHg
   * 40 bpm ≤ HR ≤ 100 bpm
   * Or considered NCS by investigators
6. Normal ECG recording on a 12-lead ECG:

   * 120 < PR < 200 ms
   * QRS < 120 ms
   * QTcf ≤ 430 ms
   * No sign of any trouble of sinusal automatism
   * Or considered NCS by investigators
7. Laboratory parameters within the normal range of the laboratory (haematological, blood chemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator
8. Normal dietary habits
9. Signing a written informed consent prior to selection

Exclusion Criteria:

1. Any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, haematological, neurologic, psychiatric, systemic, infectious or ocular disease
2. Frequent headaches and / or migraine, recurrent nausea and / or vomiting
3. Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in SBP or DBP equal to or greater than 20 mmHg within two minutes when changing from the supine to the standing position
4. Blood donation (including in the frame of a clinical trial) within 2 months before administration or apheresis within 20 days before administration
5. General anaesthesia within 3 months before administration
6. Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician (including allergy to fluorescein)
7. Inability to abstain from intensive muscular effort
8. No next of kin, easily accessible, in case of emergency
9. Any drug or herbal medicine intake (except paracetamol) during the last 14 days prior to the first administration, any over the counter medicine or vitamin during the last 7 days prior to the first administration
10. Subjects who have taken drug metabolizing enzyme inducing agents and inhibitors such as barbitals within a month prior to the first administration
11. History or presence of drug or alcohol abuse (alcohol consumption > >21 units per week)
12. Excessive consumption of beverages with xanthine bases (> 5 cups or glasses / day) and not able to stop 24h prior to admission until discharge
13. Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2
14. Major surgery (general or ocular) within 28 days prior to randomization or major surgery planned during the next 6 months
15. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development
16. Subjects within an exclusion period of a previous study or subjects who have taken any investigational product from other clinical trials within 60 days from the start of the study (from the administration of investigational product)
17. Subjects with previous participation in the current study
18. Subject under administrative or legal supervision
19. Subjects with an allergy to Fluorescein
20. History of any ocular surgery within the past 6 months prior to study participation
21. Subject who have intraocular pressure > 21 mmHg
22. Subject with acute or chronic eye problems that require eye drop at the time of screening
23. Best-corrected ETDRS visual acuity score ≤ 85 (Snellen equivalent 20/20)
24. Subject who need to wear contact lens during the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Clinical parameter: Adverse Events (AE) | During 72hours
  AEs will be coded according to the MedDRA. They will be classified into pre-defined standard categories according to chronological criteria
Local tolerance: Redness, Tingling and Other ophthalmic adverse events | During 72hours
  Redness, tingling and others should be checked

SECONDARY OUTCOMES:
Pharmacokinetic assessment: Cmax | 0hour (Pre-dose), 0.25hour, 0.5hour, 0.75hour, 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 11hour, 12hour, 24hour, 72hour
  observed maximum plasma concentration of HL217
Pharmacokinetic assessment: Tmax | 0hour (Pre-dose), 0.25hour, 0.5hour, 0.75hour, 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 11hour, 12hour, 24hour, 72hour
  first time to reach Cmax
Pharmacokinetic assessment: AUClast | 0hour (Pre-dose), 0.25hour, 0.5hour, 0.75hour, 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 11hour, 12hour, 24hour, 72hour
  area under the plasma concentration curve from administration up to the last quantifiable concentration at time 72h
Pharmacokinetic assessment: AUCinf | 0hour (Pre-dose), 0.25hour, 0.5hour, 0.75hour, 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 11hour, 12hour, 24hour, 72hour
  area under the plasma concentration-time curve from administration up to infinity with extrapolation of the terminal phase
Pharmacokinetic assessment: Kel | 0hour (Pre-dose), 0.25hour, 0.5hour, 0.75hour, 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 11hour, 12hour, 24hour, 72hour
  elimination rate constant
Pharmacokinetic assessment: T1/2 | 0hour (Pre-dose), 0.25hour, 0.5hour, 0.75hour, 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 11hour, 12hour, 24hour, 72hour
  plasma elimination half-life
Pharmacokinetic assessment: %AUCextra | 0hour (Pre-dose), 0.25hour, 0.5hour, 0.75hour, 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 11hour, 12hour, 24hour, 72hour
  percentage of extrapolated AUCinf
Pharmacokinetic assessment: Cl/F | 0hour (Pre-dose), 0.25hour, 0.5hour, 0.75hour, 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 11hour, 12hour, 24hour, 72hour
  clearance
Pharmacokinetic assessment: Vd/F | 0hour (Pre-dose), 0.25hour, 0.5hour, 0.75hour, 1hour, 2hour, 3hour, 4hour, 6hour, 8hour, 11hour, 12hour, 24hour, 72hour
  volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: David Bell, Principal Investigator — BioKinetic Europe